CLINICAL TRIAL: NCT00645307
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study With an Open-Label Extension Evaluating Extended Release OROS® Paliperidone in the Prevention of Recurrence in Subjects With Schizophrenia - Open Label Phase
Brief Title: A 52 Week Open Label Extension Trial Following the Recurrence Prevention Study R076477-SCH-301 to Evaluate the Safety and Tolerability of Paliperidone ER in Subjects With Schizophrenia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR003289
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia
Keywords: paliperidone; Schizophrenia
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: Extended Release OROS® Paliperidone

SUMMARY:
The purpose of the study was an Open Label Extension to the recurrence prevention study to evaluate long-term safety and tolerability of paliperidone ER in subjects with schizophrenia.

DETAILED DESCRIPTION:
The primary objective of the open-label extension was the long-term assessment of safety and tolerability of ER OROS paliperidone 3 to 15 mg/day in subjects diagnosed with schizophrenia. In addition, the long-term efficacy and effect of ER OROS paliperidone on overall functioning and personal and social functioning, as well as quality of life, health economics, and subjective sleep measures, was explored. This open-label extension study followed a recurrence prevention study (R076477-SCH-301) that had both an open-label run-in/stabilization phase and a double-blind, placebo-controlled phase.

Open-label study drug (ER OROS paliperidone 3 mg to 15 mg/day) was administered for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who had experienced a recurrence event during the double blind phase of Study R076477-SCH-301
* Remained recurrence free until the end of the double-blind phase, or were in the run-in or stabilization phases when the study was terminated
* Who signed the informed consent for the open-label extension
* And who the investigator agreed that open-label treatment was in the best interest of the subject were eligible to participate in the open-label extension

Exclusion Criteria:

* Not eligible to enter the open-label phase if believed to be at significant risk for suicidal or violent behavior during the open-label extension trial
* Were pregnant or had received an injection of a depot antipsychotic since entry into the preceding double-blind phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2004-05; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Long-term assessment of safety and tolerability of ER OROS paliperidone 3 to 15 mg/day in subjects diagnosed with schizophrenia

SECONDARY OUTCOMES:
Long-term efficacy and effect of ER OROS paliperidone on overall functioning and personal and social functioning, quality of life, health economics, and subjective sleep measures

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study With an Open-Label Extension Evaluating Extended Release OROS® Paliperidone in the Prevention of Recurrence in Subjects With Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=520&filename=CR003289_CSR.pdf